CLINICAL TRIAL: NCT01563224
Title: GABA-B Receptor Function in Healthy Volunteers: a Pilot, Double Blind Crossover Study of the Effects of 2 Doses of Baclofen and Placebo on Objective and Subjective Measurements of Brain Function
Brief Title: GABA-B Receptor Function in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NOAA/001/2011
Record Dates: First submitted 2012-02-13; First posted 2012-03-26 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2014-09

CONDITIONS: No Condition; Brain GABA-B Function
Keywords: GABA-B
MeSH Terms: interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- single group, crossover, 3 interventions (Experimental)
  Interventions: Drug: Baclofen 10mg; Drug: Baclofen 60mg; Drug: placebo

INTERVENTIONS:
Drug: Baclofen 10mg — Baclofen 10mg single dose po
Drug: Baclofen 60mg — Baclofen 60mg single dose po
Drug: placebo — placebo

SUMMARY:
There are several developing lines of evidence suggesting that brain receptors called GABA-B receptors play a significant role in addiction and its treatment. The investigators wish to examine the sensitivity of brain GABA-B receptors in alcohol and opiate addicts as part of the investigators MRC programme of research in neurotransmitters in alcohol and opiate addiction (NOAA). In this present study the investigators will give 2 different single doses of a drug called baclofen, and a placebo, to 8 healthy male volunteers. This drug affects GABA-B receptors in the central nervous system and is licensed for the treatment of spasticity in people with eg spinal injuries; the investigators are interested in its effects on brain GABA-B receptors. The investigators will measure EEG (brainwaves), eye movements, blood pressure and heart rate, motor co-ordination and subjective effects and also blood levels of the drug in the investigators volunteers before and at intervals after dosing. The investigators will use a double-blind randomised design to minimise expectation effects. The study will provide information on timing and magnitude of effects of baclofen on brain function in healthy subjects so that the investigators can optimise selection and timing of functional measures in future studies of addicts.

DETAILED DESCRIPTION:
After informed consent and screening participants will attend for 3 study days. On each of these there will be a set of baseline measurements including EEG, saccadic eye movements, vital signs, motor co-ordination task, subjective visual analogue ratings and questionnaires and blood sample. After dosing these measurements will be repeated at intervals during the day up to 6 hours after dosing. Participants will be allowed home after a health check.

ELIGIBILITY:
Inclusion Criteria:

* Currently healthy
* Non-smoker
* Willing to comply with protocol
* Excellent understanding of English (for questionnaires)
* Alcohol consumption between 1 and 28 units/week

Exclusion Criteria:

* Current or past history of psychiatric or substance use disorder

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
EEG spectral power in theta band | Change from baseline to 4 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lingford-Hughes, MRCPsych PhD, Principal Investigator — Imperial College London
Locations (1):
- Neuropsychopharmacology, Imperial College, London, United Kingdom